CLINICAL TRIAL: NCT01542281
Title: Improving Outcomes in Patients With Hepatobiliary Cancers With a Nutritional and Physical Conditioning Pre-habilitation Program
Brief Title: Pre-habilitation to Improve Outcomes in Patients Undergoing Liver Resection for Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Prosanto Chaudhury, HPB and Transplant Surgeon, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BMA-10-375
Record Dates: First submitted 2012-02-16; First posted 2012-03-02 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-02

CONDITIONS: Colorectal Neoplasm; Biliary Tract Neoplasm; Liver Neoplasm
Keywords: liver resection; hepatectomy; pre-habilitation
MeSH Terms: conditions — Colorectal Neoplasms; Biliary Tract Neoplasms; Liver Neoplasms | interventions — Whey Proteins; Dietary Supplements; Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutritional supplementation and prehab (Experimental): The first group (pre-hab) will receive both nutritional supplementation and a prehabilitation program.
  Interventions: Dietary Supplement: Whey protein and dietary supplements
- Prehab exercise (Active Comparator)
  Interventions: Other: prehab exercise

INTERVENTIONS:
Dietary Supplement: Whey protein and dietary supplements — Whey protein and dietary supplements in addition to pre-hab exercise
  Arms: Nutritional supplementation and prehab
Other: prehab exercise — minimum 4 weeks and maximum 8 weeks; 3 times a week
  Other Names: weight training , walking, cycling etc.
  Arms: Prehab exercise

SUMMARY:
1. To determine whether a combined nutritional support program and exercise-based prehabilitation is superior to nutritional support alone in increasing functional recovery and reducing post-operative morbidity after surgery for HPB malignancy.
2. To understand which measures of immediate surgical recovery are sensitive to prehabilitation interventions and predict change in later outcome measures.

DETAILED DESCRIPTION:
Patients scheduled for elective liver resection be will be approached andrandomized to one of two groups using a computer generated block randomisation scheme. The first group (pre-hab) will receive both nutritional supplementation and a prehabilitation program as outlined below. The second group (nutrition) will receive only nutritional supplementation. Both groups will be given a post-operative exercise program.

Once randomized, the subjects will be called by the research co-ordinator and an appointment will be made for the initial assessment. After the study is explained and consent obtained, subjects will be tested on 6MWT, followed by a 30 minute rest period during which various questionnaires assessing physical activity, quality of life, fatigue and nutritional status will be completed with the aid of the coordinator.

The prehabilitation program will last a minimum of four weeks and a maximum of 8 weeks.

Surgery will be performed by one of the HPB surgeons at the McGill University Health Center. Surgical approach, including laparoscopic or open surgery will be at the discretion of the surgeon. Perioperative care will follow an Enhanced Recovery After Surgery (ERAS)-based clinical care pathway27, 28, a fast-track care plan including patient education, afferent neural blockade, multimodal analgesia, early oral intake and mobilization, early removal of catheters and drains, and a planned 6-8 day hospital admission. This pathway has already been implemented at the Royal Victoria Hospital as part of standard patient care.

ELIGIBILITY:
Inclusion Criteria:

* Subjects eligible to enter the prehabilitation program will include those aged 18 and above and referred electively for resection of malignancies.

Exclusion Criteria:

* Excluded will be persons with American Society of Anesthesiologists (ASA) health status class 4-5 or co-morbid medical, physical and mental conditions (e.g. dementia, disabling orthopedic and neuromuscular disease, psychosis), cardiac abnormalities, severe end-organ disease such as cardiac failure, COPD, and hepatic failure (ALT and AST >50% over the normal range), and sepsis), morbid obesity (BMI >40), anemia (hematocrit < 30 %) and other conditions interfering with the ability to perform exercise at home or to complete the testing procedures.
* Patients will be excluded if they have poor English or French comprehension.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Change in six minute walk test | 8 weeks pre-op and 1 week pre-op
  The primary outcome is patient-relevant, functional walking capacity as measured by the six-minute walk test (6MWT). The 6MWT evaluates the ability of an individual to maintain a moderate level of physical activity over a time period reflective of the activities of daily living

SECONDARY OUTCOMES:
post-operative complications | 30 days
  Postoperative complications including surgical site infection, other infectious complications (such as pneumonia, urinary tract infection, line sepsis), bile leak, hemmorrhage, deep vein thrombosis, etc., will be recorded and scored using the Clavien Classification.
Health-related quality of life (HRQL) | 8 and 1 week pre-operatively, 4 and 8 weeks post-operatively
  Health-related quality of life (HRQL) as measured by the acute (1 week recall period) SF-36 health survey. The SF-36 is the most widely used HRQL measure and has been validated for surgical population; Canadian norms are also available.
Physical activity level | 8 and 1 weeks pre-operatively, 4 and 8 weeks post-operatively
  Physical activity level will be measured through the Community Health Activities Model Program for Seniors (CHAMPS) questionnaire. The CHAMPS is a self-reported measure of physical activity, comprising 41 activities evaluated according to the total number of hours done during an average week.
Depression and anxiety | 8 and 1 weeks pre-operatively, 4 and 8 weeks post-operatively
  Depression and anxiety will be assessed by The Hospital Anxiety and Depression Scale (HADS), a 14-question measure with seven items each for depression and anxiety. HADS generates separate scores for anxiety and depression as well as a combined score of psychological distress.
Fatigue | 8 and 1 weeks pre-operatively, 4 and 8 weeks post-operatively
  Fatigue will be assessed using a visual analog scale (1-10) and the Brief Fatigue Inventory (BFI). The BFI assesses the level of fatigue and its impact on activities of daily living44
Nutritional status | 8 and 1 weeks pre-operatively, 4 and 8 weeks post-operatively
  Nutritional status will be assessed through subjective and objective evaluations.Body composition will be measured by bioimpedance assay.Assessment of usual food intake will be performed using the 3-day, 24-hour food recall method. The scored Patient Generated Subjective Global Assessment (sPG-SGA) is a validated questionnaire used to assess the nutritional and functional status of cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Prosanto Chaudhury, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Royal Victoria Hospital, Montreal, Quebec, Canada